CLINICAL TRIAL: NCT04021602
Title: Diabetes Prevention Program Feasibility Study of Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Ascension Via Christi Hospitals Wichita, Inc. (Other); Kearny County Hospital (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lisette Jacobson, Assistant Professor, Preventive Medicine, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KU-VC1752; 1K01DK113048-01A1 (NIH)
Record Dates: First submitted 2019-06-12; First posted 2019-07-16 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy; Overweight and Obesity
Keywords: diabetes prevention program; breastfeeding; prediabetes
MeSH Terms: conditions — Overweight; Obesity; Breast Feeding; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care (Active Comparator): Patients randomized to Tx1 will receive education in both the Diabetes Prevention Program (DPP) and in Breastfeeding. At baseline, this includes 16 DPP sessions (core curriculum), one 2-hour breastfeeding session, and participation in a professional peer support group. The 2-hour breastfeeding session is pre-recorded into four (4) 30-minute sessions and archived on a secure, private Facebook group. Participants will have access to all four breastfeeding sessions by week 24 of pregnancy and they need to complete all sessions by week 30 of pregnancy. At delivery, the patient will receive usual lactation support in the hospital, additional breastfeeding assessment and support (at day 3, day 10, week 3 and week 6), followed by 6 DPP sessions (post-core curriculum).
  Interventions: Behavioral: Diabetes Prevention Program; Behavioral: Breastfeeding Education; Behavioral: Usual Care
- Intervention 2 (Tx2) - DPP Only + Usual Care (Active Comparator): Patients randomized to Tx2 will receive education in only the Diabetes Prevention Program. At baseline, this includes 16 DPP sessions (core curriculum). At delivery, the patient will receive usual lactation support in the hospital, followed by 6 DPP sessions (post-core curriculum).
  Interventions: Behavioral: Diabetes Prevention Program; Behavioral: Usual Care
- Intervention 3 (Tx3) - Usual Care Only (Placebo Comparator): Patients randomized to Tx3 will receive only usual standard of care. At baseline, the patient will receive only regular prenatal care provided by their physician. At delivery, the patient will receive standard of care breastfeeding support provided by the hospital.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — Phase 1 (core curriculum) of the Diabetes Prevention Program consists of 16 sessions and will take place during Week 18 of pregnancy through Week 33. Participants will receive the DPP curriculum via virtual pre-recorded sessions to which participants will have access. A research coordinator will follow up with each study participant by phone once weekly. If participants do not make adequate progress, the coordinator will assess how much extra time the participant will need to complete each session and will work with the participant if needed. Phase 2 (post-core curriculum) consists of 6 sessions and will be completed after delivery, between Week 6 and Week 20 postpartum. Participants will re-engage into the DPP with an orientation session at Week 6 postpartum. The same session completion format and procedure for inadequate progress will be followed as during pregnancy.
  Arms: Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care; Intervention 2 (Tx2) - DPP Only + Usual Care
Behavioral: Breastfeeding Education — Participants will receive a 2-hour session on breastfeeding and participate in a professional peer support group. The breastfeeding session is between Week 20 and Week 36 of pregnancy and will be taught by an International Board Certified Lactation Consultant (IBCLC). Participants will be provided with a breastfeeding assessment at Days 3 and 10; Week 3 and 6; and Months 2, 3, and 6 postpartum.
  Arms: Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care
Behavioral: Usual Care — Participants will receive regular prenatal care provided by their physician. At delivery, all participants will receive some type of lactation support in the hospital.

SUMMARY:
The purpose of this study is to learn about the impact of the Diabetes Prevention Program (DPP) coupled with intensive breastfeeding support to help overweight or obese pregnant women lose weight postpartum, improve their blood sugars and blood pressure, and increase duration of breastfeeding their infant.

DETAILED DESCRIPTION:
This pilot randomized controlled trial seeks to determine the feasibility and efficacy of a combined breastfeeding, DPP-based program in a cohort of overweight/obese women to be followed during pregnancy through 6 months postpartum. The pilot trial will have three study arms: DPP + breastfeeding (Tx1), DPP only (Tx2), and usual care (Tx3). Specific aims are: 1) To test the efficacy of Tx1 to improve 6-month postpartum weight loss among women with a BMI >/= 25. 2) To test the efficacy of Tx1 to improve 6-month postpartum mean blood glucose (HbA1c) and mean arterial blood pressure among women with a BMI >/= 25. 3) To test the efficacy of Tx1 to increase any breastfeeding through 6 months postpartum among women with a BMI >/= 25.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant, 1st trimester or early 2nd trimester
* Interested in breastfeeding
* BMI >/= 25 and <35
* Able to read and understand English
* Able to learn and use Facebook
* Able to learn and use Skype, FaceTime or Zoom for virtual meetings
* Must have a cell phone

Exclusion Criteria:

* Pregnancy complications that require emergency care
* Thyroid disease
* Multiple gestation
* Substance abuse within last 3 years
* ART (Assisted Reproductive Technology) pregnancy
* Current smoker
* Prior bariatric surgery
* In weight-loss program within 3 months of conception
* BMI >/= 35
* Unable to attend intervention / follow-up visits
* Unwilling to self-monitor data collection
* Unable to complete intervention
* Presence of any condition that limits walking
* Presence of any condition that limits following diet recommendations
* Pregnancies complicated with fetuses diagnosed with lethal malformations / conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Kearny County Hospital, Lakin, Kansas
  - Via Christi Maternal Fetal Medicine Clinic, Wichita, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jacobson LT, Bakhache N, Dowling J, Okut H, Zackula R, Robbins DC, Stern JE, Grainger DA, Befort C. Electronic Monitoring of Mom's Schedule (eMOMSTM): A Qualitative Study of Experiences in a Lifestyle Change Program with Lactation Support. Am J Health Promot. 2023 Sep;37(7):953-963. doi: 10.1177/08901171231189540. Epub 2023 Jul 18. PMID 37461383

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care: Participants randomized to Tx1 will receive education in the Diabetes Prevention Program (DPP) and in Breastfeeding. At baseline, this includes 16 DPP sessions, one breastfeeding session, and participation in a professional peer support group. At delivery, the patient will receive usual lactation support in the hospital, additional breastfeeding assessment and support, followed by 6 DPP sessions.
  DPP: Phase 1 consists of 16 sessions during Week 18 of pregnancy through Week 33. Participants will receive the DPP curriculum via virtual pre-recorded sessions. Phase 2 (post-core) consists of 6 sessions and will be completed after delivery, between Week 6 and Week 20 postpartum. Participants will re-engage into the DPP with an orientation session at Week 6 postpartum.
  Breastfeeding: Participants will receive a 2-hour session on breastfeeding and participate in a professional peer support group. The breastfeeding session is between Week 20 and Week 36 of pregnancy and will be taught by an International Board Certified Lactation Consultant (IBCLC). Participants will be provided with a breastfeeding assessment at Days 3 and 10; Week 3 and 6; and Months 2, 3, and 6 postpartum.
  Usual Care: Participants will receive regular prenatal care provided by their physician. At delivery, all participants will receive some type of lactation support in the hospital.
- Intervention 2 (Tx2) - DPP Only + Usual Care: Patients randomized to Tx2 will receive education in only the Diabetes Prevention Program. At baseline, this includes 16 DPP sessions. At delivery, the patient will receive usual lactation support in the hospital, followed by 6 DPP sessions.
  DPP: Phase 1 consists of 16 sessions during Week 18 of pregnancy through Week 33. Participants will receive the DPP curriculum via virtual pre-recorded sessions. Phase 2 (post-core) consists of 6 sessions and will be completed after delivery, between Week 6 and Week 20 postpartum. Participants will re-engage into the DPP with an orientation session at Week 6 postpartum.
  Usual Care: Participants will receive regular prenatal care provided by their physician. At delivery, all participants will receive some type of lactation support in the hospital.
Period: Overall Study
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Started | 9 | 14 | 12
Completed | 5 | 11 | 10
Not Completed | 4 | 3 | 2
Not completed — Lost to Follow-up | 3 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only | Total
Number analyzed (Participants) | 9 | 14 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (7.4) | 27.1 (5.2) | 27.6 (5.4) | 27.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 12 | 35
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: Non-Hispanic White | 7 | 8 | 8 | 23
  Ethnicity/Race: Hispanic | 1 | 2 | 2 | 5
  Ethnicity/Race: Non-Hispanic Black | 0 | 3 | 1 | 4
  Ethnicity/Race: Other | 1 | 1 | 1 | 3
Location [Count of Participants; unit: Participants]
  Rural | 0 | 1 | 2 | 3
  Urban | 9 | 13 | 10 | 32
Highest Level of Education Completed [Count of Participants; unit: Participants]
  Some high school | 1 | 2 | 0 | 3
  Graduated from high school | 3 | 3 | 0 | 6
  Some college or associate's degree | 3 | 6 | 6 | 15
  Graduated with a bachelor's degree | 2 | 3 | 5 | 10
  Advanced degree (e.g. Masters, PhD, MD, JD) | 0 | 0 | 1 | 1
Gross yearly total household income before taxes during the last 12 months before current pregnancy [Count of Participants; unit: Participants]
  $9,999 or less | 1 | 4 | 4 | 9
  $10,000 to $24,999 | 1 | 3 | 0 | 4
  $25,000 to $49,999 | 4 | 3 | 2 | 9
  $50,000 to $74,999 | 2 | 1 | 2 | 5
  $75,000 or more | 1 | 3 | 4 | 8
Currently have health insurance [Count of Participants; unit: Participants]
  Yes | 9 | 14 | 12 | 35
  No | 0 | 0 | 0 | 0
WIC participation during pregnancy [Count of Participants; unit: Participants]
  Yes | 3 | 3 | 1 | 7
  No | 6 | 11 | 11 | 28
Reported immediate biological family member ever diagnosed with or treated for diabetes [Count of Participants; unit: Participants] — Immediate biological family member is defined/described as mother, father, brother, and/or sister.
  Participants
    Yes | 5 | 5 | 4 | 14
    No | 4 | 9 | 8 | 21
Pregnancy trimester at study entry [Count of Participants; unit: Participants]
  1st trimester | 4 | 9 | 8 | 21
  2nd trimester | 5 | 5 | 4 | 14
  3rd trimester | 0 | 0 | 0 | 0
Number of live births (not including current pregnancy) [Count of Participants; unit: Participants]
  None | 2 | 6 | 6 | 14
  1 birth | 2 | 4 | 2 | 8
  2 births | 2 | 2 | 2 | 6
  3 births | 1 | 0 | 1 | 2
  4 or more births | 2 | 2 | 1 | 5
Number of stillbirths [Count of Participants; unit: Participants]
  None | 7 | 12 | 12 | 31
  One | 1 | 1 | 0 | 2
  Did not answer | 1 | 1 | 0 | 2
Had a preterm delivery (baby was born before 37 weeks of pregnancy) [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 0 | 3
  No | 7 | 13 | 12 | 32
Type of diabetes (if diagnosed with pregestational diabetes) [Count of Participants; unit: Participants]
  Type 1 diabetes | 0 | 1 | 0 | 1
  Type 2 diabetes | 0 | 1 | 0 | 1
  Not diagnosed with pregestational diabetes | 9 | 12 | 12 | 33
Smoking status [Count of Participants; unit: Participants]
  Not currently smoking | 9 | 14 | 12 | 35
  Currently smoking | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: The study team will measure maternal weight at baseline, at delivery, and weekly during the postpartum period to allow for meaningful comparisons of weight change among study arms.
Time Frame: At baseline and at delivery through 6 months postpartum
Population: We were unable to collect weight at certain time points for some participants.
Measure: Median (Inter-Quartile Range); unit: kgs
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 8
kgs
  Baseline - delivery (GWG): number analyzed (Participants) | 4 | 9 | 6
  Baseline - delivery (GWG) | 7.5 [5.7 to 10.2] | 13.4 [9.4 to 18.3] | 18.2 [8.6 to 22.8]
  Delivery - 6 month postpartum: number analyzed (Participants) | 4 | 9 | 6
  Delivery - 6 month postpartum | -5.6 [-6.4 to -3.1] | -12.3 [-13.7 to -7.9] | -11.2 [-15.5 to -4.3]
  Baseline - 6 month postpartum | 4.1 [2.0 to 5.7] | 3.5 [3.4 to 7.2] | 5.9 [4.0 to 10.3]

2. Primary Outcome: Change in HbA1c
Description: The study team will measure mean blood glucose at baseline and at 6 months postpartum.
Time Frame: At baseline and at 6 months postpartum
Population: We were unable to collect HbA1c at certain time points for some participants.
Measure: Median (Inter-Quartile Range); unit: mmol/mol
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 9
mmol/mol
  Baseline: number analyzed (Participants) | 3 | 11 | 9
  Baseline | 5.2 [4.7 to 5.4] | 5.2 [4.8 to 5.8] | 5.0 [5.0 to 5.2]
  6 months: number analyzed (Participants) | 5 | 11 | 8
  6 months | 5.3 [5.2 to 5.4] | 5.4 [5.0 to 5.7] | 5.1 [5.0 to 5.2]

3. Primary Outcome: Change in Arterial Blood Pressure
Description: The study team will measure mean arterial blood pressure at baseline and at 6 months postpartum.
Time Frame: At baseline, at delivery, and at 6 months postpartum
Population: We were unable to collect arterial blood pressure at certain time points for some participants.
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
mmHg
  Baseline | 85.0 [82.0 to 85.3] | 90.7 [77.7 to 94.0] | 89.7 [86.7 to 95.3]
  6 months: number analyzed (Participants) | 5 | 11 | 8
  6 months | 92.7 [87.3 to 94.0] | 91.3 [81.3 to 98.7] | 90.8 [85.0 to 95.0]

4. Primary Outcome: Duration of Breastfeeding
Description: The study team will measure duration of breastfeeding from delivery through 6 months postpartum.
Time Frame: At delivery through 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
Participants
  10 days: Still Breastfeeding | 4 | 7 | 6
  10 days: No longer breastfeeding | 1 | 4 | 4
  6 weeks: Still Breastfeeding | 3 | 4 | 4
  6 weeks: No longer breastfeeding | 2 | 7 | 6
  3 months: Still Breastfeeding | 3 | 3 | 3
  3 months: No longer breastfeeding | 2 | 8 | 7
  6 months: Still Breastfeeding | 2 | 2 | 1
  6 months: No longer breastfeeding | 3 | 9 | 9

5. Secondary Outcome: Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF, Survey)
Description: To assess levels of self-efficacy. Survey consists of 14 items. All items are preceded by the phrase "I can always" and are anchored with a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. All items are presented positively, and scores are summed to produce a range from 14 to 70, with higher scores indicating higher levels of breastfeeding self-efficacy.
Time Frame: At baseline and at 6 months postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
score on a scale
  Baseline | 33.0 [28.0 to 50.0] | 35.0 [20.0 to 44.0] | 41.0 [32.0 to 49.0]
  6 months | 49.0 [26.0 to 52.0] | 52.0 [27.0 to 70.0] | 62.5 [30.0 to 65.0]

6. Secondary Outcome: Kaiser Physical Activity Survey (KPAS, Weighted Total)
Description: To assess multiple domains of physical activity and total physical activity before and after pregnancy. Survey consists of 38 items; 4 domains: household and family care activities, occupational activities, active living habits, participation in sports/exercise. Activity indices were created for each domain of activity by summing the domain-specific categorical responses and dividing by the number of items, giving an average value that ranged from 1 to 5 (scores ranged from 1 for "never" or "none" to 5 for "always" or "more than once a week" in each physical activity domain). Higher scores indicate greater overall activity levels. Total activity index is calculated as the sum of all four indices: Total activity = (household/caregiving index*0.25 + occupational index*0.25 + active living index*0.25 + sports/exercise index*0.25) * 4. The total activity score has a potential range of 4 - 20 with a mean of 10.42 (SD=2.00). A higher total activity score indicates a greater activity level.
Time Frame: At baseline and at 6 months postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
score on a scale
  Baseline | 12.1 [12.0 to 12.9] | 10.1 [9.3 to 11.1] | 10.6 [9.7 to 11.3]
  6 months | 12.4 [11.7 to 15.1] | 12.2 [10 to 13.4] | 10.6 [9.7 to 11.3]

7. Secondary Outcome: Fruit & Vegetable Intake Screener (EATS)
Description: To assess intake of fruits and vegetables before and after pregnancy. Survey consists of 10 items; with portion-size questions. Each question has two parts, asking over the last month how often a particular item was consumed (i.e.: never, 1-3x/mo, 1-2x/wk, etc.) and how much was usually consumed (i.e.: <3/4cup, 3/4 to 1 1/4 cup, >2 cups, etc.). Frequency is scored from 0.0-5.0, with 0 meaning never, and 5.0 meaning 5 or more servings per day.
Time Frame: At baseline and at 6 months postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
score on a scale
  Baseline | 1.6 [1.2 to 2.8] | 1.8 [1.1 to 2.5] | 1.9 [1.3 to 2.7]
  6 months | 1.9 [1.4 to 2.2] | 1.8 [1.3 to 2.7] | 3.1 [1.9 to 4.5]

8. Secondary Outcome: Edinburgh Postnatal Depression Scale (EPDS)
Description: To assess levels of depression during the postpartum period. Survey consists of 10 items. Questions 1, 2, & 4 are scored 0, 1, 2 or 3 with top box scored as 0 and the bottom box scored as 3. Questions 3, 5--10 are reverse scored, with the top box scored as a 3 and the bottom box scored as 0. Maximum score is 30. A score of 10 or higher generally indicates a potential need for further assessment regarding possible depression, while scores above 12 or 13 may suggest a higher likelihood of depression requiring medical attention. Participants with a score of 10 or greater will be referred to their healthcare provider for follow up.
Time Frame: Postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
Number analyzed (Participants) | 5 | 11 | 10
score on a scale
  Week 3 | 7 [6 to 8] | 6 [2 to 6] | 5 [4 to 9]
  Week 6 | 7.5 [6.5 to 10] | 6 [0 to 9] | 4 [1.5 to 4]
  Week 12 | 9 [6.5 to 13.5] | 6 [0 to 7] | 3 [1 to 5]
  Month 6 | 7.5 [5.5 to 9.5] | 4 [1 to 9] | 3 [1 to 4]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through 6 months postpartum follow up.
Arm/Group | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care | Intervention 2 (Tx2) - DPP Only + Usual Care | Intervention 3 (Tx3) - Usual Care Only
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/14 | 1/12
Other Adverse Events (participants affected / at risk) | 0/9 | 0/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention 1 (Tx1) - DPP + Breastfeeding + Usual Care (N=9) | Intervention 2 (Tx2) - DPP Only + Usual Care (N=14) | Intervention 3 (Tx3) - Usual Care Only (N=12)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 1 (1) — The miscarriage was unrelated to the study or any study activities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT04021602/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT04021602/ICF_001.pdf